CLINICAL TRIAL: NCT06178458
Title: Prediction of Pain Score and Opioid Consumption of Index Cesarean Delivery From Pain Score and Opioid Consumption of Previous Cesarean Delivery: A Retrospective Study
Brief Title: Pain Score and Opioid Consumption of Index and Previous Cesarean Delivery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sasikaan Nimmaanrat, Associate Professor, Prince of Songkla University
Other Study IDs: 66-348-8-1
Record Dates: First submitted 2023-12-11; First posted 2023-12-21 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Pain; Postoperative
Keywords: cesarean delivery; opioid consumption; pain score
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention — To collect data of pain score and opioid consumption of index and previous cesarean delivery

SUMMARY:
Postoperative pain after cesarean delivery is common and affects on both mothers and children.

The goals of this retrospective observational study aim to predict pain score and opioid consumption of index cesarean delivery from pain score and opioid consumption of previous cesarean delivery.

DETAILED DESCRIPTION:
The authors will review the medical records of recruited participants for demographic data as well as pain scores and opioid consumption of index cesarean delivery and previous cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had at least 2 cesarean deliveries
* Patients received spinal anesthesia and intrathecal morphine for cesarean delivery
* Patients received postoperative pain control as per standard protocol

Exclusion Criteria:

* Patients with chronic pain prior to cesarean delivery
* Unable to give pain score
* Receiving general anesthesia for cesarean delivery
* Receiving postoperative pain control beyond the standard protocol
* Patients with multiple pregnancy, placenta abruption, placenta accrete, postpartum hemorrhage
* Patients with psychotic disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female because only females can have cesarean delivery
Study Population: Patients scheduled for cesarean delivery under spinal anesthesia with intrathecal morphine.
Sampling Method: Probability Sample
Enrollment: 416 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prediction of pain score after cesarean delivery | January 2024 - December 2025
  To predict pain score of index cesarean delivery from previous cesarean delivery using pain score measured by verbal numerical rating scale (VNRS) ranging from 0 (no pain) to 10 (worst pain imaginable).

SECONDARY OUTCOMES:
Prediction of opioid consumption after cesarean delivery | January 2024 - December 2025
  To predict opioid consumption of index cesarean delivery from previous cesarean delivery based on 1. number and percentage of patients who required opioid for controlling postoperative pain, 2. MME (milligram morphine equivalent) per total patients and 3. MME per patients who received opioid

CONTACTS AND LOCATIONS:
Overall Officials: Boonsin Tangtrakulwanich, MD, Study Chair — Prince of Songkla University

IPD SHARING:
Plan to Share IPD: Undecided
IPD to be shared upon request.